CLINICAL TRIAL: NCT01560078
Title: Evaluation of Efficacy of Thrice Weekly DOTS Regimen in Tubercular Pleural Effusion at 6 Months
Brief Title: Efficacy Study of Thrice Weekly Directly Observed Treatment Short-Course Regimen in Tubercular Pleural Effusion
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Sri Venkateswara Institute of Medical Sciences University (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head of Department, All India Institute of Medical Sciences
Other Study IDs: T-18012/2/2005-TB/CCD
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Tuberculosis; Pleural Effusion
Keywords: Tuberculosis; Pleural effusion; Category 3
MeSH Terms: conditions — Tuberculosis; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tubercular pleural effusion is the second most common form of extrapulmonary tuberculosis (EPTB) seen in clinical practice after tuberculosis (TB) lymphadenitis. It is common that after complete treatment of the patient with tubercular pleural effusion with six months of the short-course chemotherapy under Directly Observed Treatment Short-Course (DOTS), pleural effusion has not resolved completely. In these cases treatment need to be extended for one or two more months by giving extension pouches.

Since DOTS does not recommend demonstration of complete resolution of tubercular pleural effusion at the end of treatment completion, there is paucity of data in terms of the patients declared cure for the sputum negative pulmonary and extra-pulmonary TB as such which includes TB pleural effusion as well. This project aims to look into the patient characteristics, treatment outcome, and compute the number of cases which require an extended regimen and to what extent is the pleural effusion persistent at the end of six months of standard DOTS therapy.

DETAILED DESCRIPTION:
India's Revised National Tuberculosis Control Programme (RNTCP), based on Directly Observed Treatment Short-Course (DOTS) strategy, began as a pilot project in 1993 and was launched as a national program in 1997. Three categories of treatment were recommended based on disease characteristics. Category III regimen comprised of thrice-weekly isoniazid, rifampicin and pyrazinamide in the intensive phase; with isoniazid and rifampicin in the continuation phase. This regimen was recommended for sputum smear negative and extrapulmonary tuberculosis (TB) patients who were not seriously ill. The omission of ethambutol in non-cavitary, smear-negative pulmonary TB patients who were known to be human immunodeficiency virus (HIV) negative was endorsed by the World Health Organization (WHO) guidelines. However, in view of high level of initial resistance to isoniazid in many areas, recent guidelines recommend adding ethambutol in the intensive phase, effectively eliminating category III.

This study was designed as a multicentre, longitudinal observational study and was carried out between 2006 and 2011. Three hundred and sixty patients were planned to be enrolled across 4 centres, namely AIIMS (New Delhi), SMS Medical College (Jaipur), SVIMS (Tirupati) and BJ Medical College (Ahmedabad); i.e. 90 patients at each centre. Lost to follow-up/default rate of 12% was expected in the study. Recruitment was done from the study sites directly as well as from referrals via nearby DOTS centres, hospitals and chest clinics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral TB pleural effusion < 1500 ml

Exclusion Criteria:

* Patients < 15 years and > 65 years were excluded
* Patients with opacity greater than four intercostal spaces in the posteroanterior (PA) chest radiograph
* Bilateral pleural effusion
* Patients who were failures/defaulters/relapses (eligible for cat II as per RNTCP guidelines)
* Sputum-smear positive cases, miliary TB, moderately advanced and far advanced parenchymal involvement on chest radiograph (eligible for cat I)
* HIV positive
* Hepatitis B surface antigen (HBsAg) positive
* Diabetes mellitus
* Refusing thoracocentesis
* Evidence of empyema
* Residence outside the study area
* Refuse to give consent

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1042 patients presenting with unilateral tubercular pleural effusion who attended DOTS Centres/Chest clinics at the respective Study sites between the ages 15 and 65 years were screened for the study.351 were enrolled after 691 were excluded due to various reasons.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2006-09; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Complete resolution of pleural effusion on ultrasonogram | 6 months
  Ultrasonogram to monitor pleural fluid done at baseline,2 months, 4 months and 6 months from enrollment to monitor resolution

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD,PhD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India